CLINICAL TRIAL: NCT00952328
Title: Effect of Early Limited Formula Use on Breastfeeding Outcomes
Acronym: ELF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H49316-34032-01; 5 K12 HD052 163 Development
Record Dates: First submitted 2009-07-29; First posted 2009-08-06 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Breastfeeding
Keywords: breastfeeding outcomes; breastfeeding self-efficacy; infant weight loss
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Limited Formula (Experimental): Participants will supplement feedings with early limited formula following nursing
  Interventions: Dietary Supplement: Nutramigen infant formula
- Control (No Intervention): Participants are instructed to continue exclusively breastfeeding; no use of formula

INTERVENTIONS:
Dietary Supplement: Nutramigen infant formula — Investigators will advise mothers to supplement with 10 cc of elemental formula immediately following each breastfeeding and to discontinue formula once mature milk production begins.
  Arms: Limited Formula

SUMMARY:
The aim of this study is to conduct a pilot randomized controlled trial of the effect of early limited formula supplementation on breastfeeding-related outcomes for infants with high early weight loss. The investigators will enroll 40 exclusively breastfeeding infants at 24-48 hours of age and will randomly assign them to early limited formula supplementation following nursing (intervention group) or to no formula feeding (control group). Both groups will receive intensive lactation support. Outcome variables will include breastfeeding status on day-of-life 8, weight nadir, breastfeeding self-efficacy, maternal satisfaction, and exclusive and partial breastfeeding at 1-3 months. The hypothesis for this study is that early limited formula supplementation might help infants with early weight loss avoid eventual weight loss ≥ 10% and associated breastfeeding problems.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants (37 to 42 weeks gestation)
* Infants who have lost 5% of their birth weight at <36 hours of age

Exclusion Criteria:

* Infants who have received formula or water
* Mothers who are producing mature milk supply
* Infants receiving Level II or Level III care other than healthy term infants with routine complete blood count and blood tests pending

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Is infant receiving exclusively breast milk at 8 days of life? | 8 days following baseline

SECONDARY OUTCOMES:
Is infant receiving exclusive or partial breastfeeding at 1 month, 2 months, and 3 months? | 1-3 months following baseline

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flaherman, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Medical Center, San Francisco, California, United States